CLINICAL TRIAL: NCT00692770
Title: A Phase III Randomized, Double-blind, Placebo-controlled Study of Sorafenib as Adjuvant Treatment for Hepatocellular Carcinoma After Surgical Resection or Local Ablation.
Brief Title: Sorafenib as Adjuvant Treatment in the Prevention Of Recurrence of Hepatocellular Carcinoma (STORM)
Acronym: STORM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12414; 2008-001087-36 (EudraCT Number)
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Sorafenib; Adjuvant; Surgical resection; Ablation; Nexavar; Adjuvant therapy; Liver cancer; HCC; STORM
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Participants received 2 tablets of Sorafenib (2×200 mg) orally twice daily (BID)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)
- Placebo (Placebo Comparator): Participants received 2 tablets of placebo orally twice daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Sorafenib 400 mg twice daily (BID)
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Placebo 2 tablets twice daily (BID)
  Arms: Placebo

SUMMARY:
To evaluate efficacy and safety of sorafenib versus placebo in the adjuvant treatment of Hepatocellular Carcinoma (HCC) after potentially curative treatment (surgical resection or local ablation).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone surgical resection or local ablation (PEI or percutaneous or intraoperative RFA) for treatment of HCC with curative intent within 4 months from staging to potentially curative treatment. A maximum of 2 local ablation courses may be administered during this time period.
* At least 3 weeks (21 days) but no more than 7 weeks (49 days), from resection or last local ablation course, to CT/MRI scan date
* Male or female subjects >/= 18 years of age
* Confirmation of CR (absence of residual tumor after curative treatment), on the eligibility scan by independent radiological review.
* For subjects undergoing surgical resection pathology proven complete removal of tumor.
* Intermediate or High Risk of recurrence as assessed by tumor characteristics.
* Child-Pugh score 5 -7 points. A Child-Pugh score of 7 points is allowed only in the absence of ascites.
* ECOG Performance Status of 0.
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Recurrent HCC
* Child-Pugh score 7 points with presence of ascites.
* Low risk of recurrence after curative treatment
* History of cardiovascular disease
* History of HIV infection
* Active clinically serious infections (> grade 2 NCI-CTCAE version 3.0)
* Subjects with seizure disorder requiring medication (such as steroids or anti-epileptics)
* Subjects with evidence or history of bleeding diathesis
* Subjects undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry as defined by the signing of informed consent..
* Uncontrolled ascites (defined as not easily controlled with diuretic treatment)
* Encephalopathy
* History of GI bleeding within 30 days of randomization.
* Subjects with a history of esophageal varices bleeding which has not been followed by effective therapy and/or treatment to prevent bleeding recurrence.
* Prior anti cancer therapy for treatment of HCC (including sorafenib or any other molecular therapy) is excluded.
* Major surgery within 4 weeks of start of study as defined by the signing of informed consent, except for surgical resection or local ablation of HCC.
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry, as defined by the signing of informed consent.
* Liver transplantation, this includes patients on a transplant list with the intention to transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2008-08-15 (Actual); Primary Completion 2013-11-29 (Actual); Study Completion 2014-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (169):
- United States (24):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - New York, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Argentina (3):
  - Pilar, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Australia (5):
  - Camperdown, New South Wales
  - Randwick, New South Wales
  - Brisbane, Queensland
  - Heidelberg, Victoria
  - Melbourne, Victoria
- Austria (3):
  - Innsbruck
  - Linz
  - Vienna
- Belgium (4):
  - Bruxelles - Brussel
  - Ghent
  - Leuven
  - Liège
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - São Paulo
- Bulgaria (2):
  - Plovdiv
  - Varna
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
- Chile (2):
  - Reñaca, Región de Valparaíso
  - Santiago, Santiago Metropolitan
- China (14):
  - Guangzhou, Guangdong
  - Nanning, Guangxi
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Xi’an, Shanxi
  - Chengdu, Sichuan
  - Beijing
  - Beijng
  - Chongqing
  - Dalian
  - Hefei
  - Shanghai
  - Tianjin
- France (13):
  - Angers
  - Bondy
  - Bordeaux
  - Créteil
  - Lille
  - Lyon
  - Marseille
  - Nice
  - Paris
  - Rennes
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (14):
  - München, Bavaria
  - Regensburg, Bavaria
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Aachen, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Homburg/Saar, Saarland
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Hamburg
- Athens / Greece, Greece
- Hong Kong (3):
  - Hong Kong
  - Kwun Tong
  - Shatin
- Italy (12):
  - Bari, Apulia
  - Benevento, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Catania, Sicily
  - Palermo, Sicily
  - Padua, Veneto
- Japan (17):
  - Kashiwa-shi, Chiba
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Osakasayama-shi, Osaka
  - Suita, Osaka
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Minato-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Fukuoka
  - Kumamoto
  - Kyoto
  - Okayama
  - Osaka
  - Tokushima
- Mexico (3):
  - México, D.F., Mexico City
  - Monterrey, Nuevo León
  - México, D.F.
- Auckland, New Zealand
- Coimbra, Portugal
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (3):
  - Moscow
  - Obninsk
  - Saint Petersburg
- Singapore, Singapore
- South Korea (6):
  - Goyang-si, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Daegu
  - Jeollabuk-do
  - Seoul
- Spain (10):
  - Sabadell, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Barcelona, Catalonia
  - Majadahonda, Madrid
  - Oviedo, Principality of Asturias
  - Badajoz
  - Barcelona
  - Córdoba
  - Madrid
  - Valladolid
- Sweden (2):
  - Gothenburg
  - Stockholm
- Switzerland (2):
  - Bern
  - Zurich
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - Kaohsung
  - Tainan
  - Taipei
  - Taoyuan District
- United Kingdom (6):
  - Southampton, Hampshire
  - Birmingham, West Midlands
  - Leeds, West Yorkshire
  - London
  - Manchester
  - Newcastle upon Tyne

REFERENCES:
- [Result] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Derived] Pinyol R, Montal R, Bassaganyas L, Sia D, Takayama T, Chau GY, Mazzaferro V, Roayaie S, Lee HC, Kokudo N, Zhang Z, Torrecilla S, Moeini A, Rodriguez-Carunchio L, Gane E, Verslype C, Croitoru AE, Cillo U, de la Mata M, Lupo L, Strasser S, Park JW, Camps J, Sole M, Thung SN, Villanueva A, Pena C, Meinhardt G, Bruix J, Llovet JM. Molecular predictors of prevention of recurrence in HCC with sorafenib as adjuvant treatment and prognostic factors in the phase 3 STORM trial. Gut. 2019 Jun;68(6):1065-1075. doi: 10.1136/gutjnl-2018-316408. Epub 2018 Aug 14. PMID 30108162
- [Derived] Bouattour M, Soubrane O, de Gramont A, Faivre S. Adjuvant therapies in advanced hepatocellular carcinoma: moving forward from the STORM. Trials. 2016 Nov 25;17(1):563. doi: 10.1186/s13063-016-1675-8. PMID 27887632
- [Derived] Kudo M. Adjuvant therapy after curative treatment for hepatocellular carcinoma. Oncology. 2011;81 Suppl 1:50-5. doi: 10.1159/000333259. Epub 2011 Dec 22. PMID 22212936
- [Derived] Printz C. Clinical trials of note. Sorafenib as adjuvant treatment in the prevention of disease recurrence in patients with hepatocellular carcinoma (HCC) (STORM). Cancer. 2009 Oct 15;115(20):4646. doi: 10.1002/cncr.24673. No abstract available. PMID 19806596
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment period was between 15 August 2008 to 12 November 2010.
Pre-assignment Details: Of 1602 participants who were screened for inclusion in the study, 1114 were enrolled, and 1107 received treatment.
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Started | 556 | 558
Participants Received Treatment | 553 | 554
Completed | 0 | 0
Not Completed | 556 | 558
Not completed — Protocol Violation | 2 | 7
Not completed — Withdrawal by Subject | 97 | 36
Not completed — Adverse Event | 136 | 41
Not completed — Death | 10 | 5
Not completed — Lost to Follow-up | 7 | 3
Not completed — Non-compliant with study medication | 11 | 5
Not completed — Progression by clinical judgment | 2 | 3
Not completed — Physician decision not protocol driven | 10 | 14
Not completed — Disease progression, recurrence/relapse | 170 | 279
Not completed — Protocol driven decision point | 3 | 7
Not completed — Completed all planned assessments | 79 | 101
Not completed — Radiological and clinical progression | 8 | 8
Not completed — Clinical endpoint reached | 16 | 43
Not completed — Study terminated by sponsor | 2 | 2
Not completed — Randomized but not treated | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 556 | 558 | 1114
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (11.7) | 58.7 (12.2) | 58.4 (12.0)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 65 years | 383 | 361 | 744
  >=65 years | 173 | 197 | 370
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 97 | 202
  Male | 451 | 461 | 912

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival (RFS) by Independent Assessment
Description: Disease recurrence of HCC (intra or extra hepatic) was defined as the appearance of a new intrahepatic lesions fulfilling the American Association for the Study of Liver Diseases (AASLD) criteria of diagnosis of HCC or a new extra-hepatic lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.0. In addition to investigator assessment, all images were reviewed by an independent panel of radiologists. The calculation of the RFS was based on the independent evaluation of the scans. RFS was defined as the time from randomization to the first documented disease recurrence by independent radiological assessment or death due to any cause whichever occurred first. For subjects who had not recurred or died at the time of analysis, RFS was censored at their last date of evaluable scan before drop-out for any other reason than recurrence or death.
Time Frame: From randomization up to 4 years or until disease recurrence whichever came first
Population: Full analysis set (FAS) included participants who were randomized to study treatments.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Days | 1014 [839 to 1339] | 1026 [841 to 1185]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.258329, Log Rank — One sided P-value was stratified by region, risk of recurrence and previous curative treatment; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.78 to 1.134]

2. Secondary Outcome: Time to Recurrence (TTR) by Independent Assessment
Description: TTR was defined as the time from randomization to the first documented disease recurrence by independent radiological assessment. For subjects who had not recurred at the time of analysis, TTR was censored at their last date of evaluable scan before withdrawal for any other reason than recurrence. "NA" in the reported data indicates values could not be estimated due to censored data.
Time Frame: From randomization up to 4 years or until disease recurrence whichever came first
Population: FAS included participants who were randomized to study treatments.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Days | 1172 [924 to NA] — Value cannot be estimated due to censored data. | 1089 [923 to 1260]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.121383, Log Rank — One sided P-value was stratified by region, risk of recurrence and previous curative treatment; Hazard Ratio (HR) = 0.891, 95% CI 2-sided [0.735 to 1.081]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to date of death due to any cause. OS for subjects alive at the time of analysis was censored at their last date of contact. "NA" in the reported data indicates values could not be estimated due to censored data.
Time Frame: From randomization of the first subject until 4 years later.
Population: FAS included participants who were randomized to study treatments.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Days | NA [NA to NA] — "NA" in the reported data indicates values could not be estimated due to censored data. | NA [NA to NA] — "NA" in the reported data indicates values could not be estimated due to censored data.
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; p = 0.484742, Log Rank — One-sided P-value was stratified by region, risk of recurrence and previous curative treatment; Hazard Ratio (HR) = 0.995, 95% CI 2-sided [0.761 to 1.3]

4. Other Pre Specified Outcome: Patient Reported Outcomes: Euroqol-5 Dimensions (EQ-5D) - Index Score
Description: The EQ-5D is a generic quality of life preference based on a validated instrument used in cancer and in general population, with 2 parts: Index and Visual Analogue Scale. The EQ-5D Index is a descriptive system of the following health dimensions: mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression. Subjects were asked to choose any one of the 3 response levels for each dimension: no problems, some problems, and severe problems. The 5 health dimensions were summarized into a single score, the EQ-5D Index score which ranged from -0.59 to 1 with higher scores representing better health states (0=death, 1= perfect health, and -0.59=a health state worse than death). A change of at least 0.10 to 0.12 points was considered a minimally important difference using Eastern Cooperative Oncology Group Performance Status as the anchor. The results on the Analysis of covariance of timeadjusted Area under curve for the EQ-5D index score were reported.
Time Frame: Cycle (C) Day (D)1, C2D1, C3D1 and subsequent cycles up to C18, end of intervention visit
Population: FAS included participants who were randomized to study treatments.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Unit on a scale | 0.827 [0.804 to 0.85] | 0.866 [0.843 to 0.888]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; An analysis of covariance (ANCOVA) model was used to estimate the mean difference in the timeadjusted Area Under Curve (AUC) between the two treatment groups, with covariates for baseline scores and stratification factors. To test the treatment effect, a mixed linear model (random coefficient model) was used for the EQ-5D index score. Statistical tests were performed with a 2 sided type I error of 5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [0.025 to 0.052]

5. Other Pre Specified Outcome: Patient Reported Outcomes: Euroqol-5 Dimensions (EQ-5D) - Visual Analogue Scale (VAS) Score
Description: The EQ-5D is a generic quality of life preference based on a validated instrument used in cancer and in general population, with 2 parts: Index and Visual Analogue Scale. The EQ-5D VAS is a measure that represents health status as a single value. It is a 20-centimetre vertical graduated visual analogue scale with scores that ranged from 0 (worst imaginable health state) to 100 (best imaginable health state). The respondent rated his/her current health state by drawing a line from the box marked 'your own health state today' to the appropriate point on the EQ-5D VAS. A 3-digit number (including leading zeros) was read off the scale from the point where the respondent's line crossed the scale, which was the EQ-5D VAS score. A change of at least 7 points on the VAS was considered as minimally important. The results on the ANCOVA analysis of time-adjusted AUC for the EQ-5D VAS score were reported.
Time Frame: Cycle (C) Day (D)1, C2D1, C3D1 and subsequent cycles up to C18, end of intervention visit
Population: FAS included participants who were randomized to study treatments.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Unit on a scale | 77.203 [75.184 to 79.223] | 80.181 [78.212 to 82.151]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; An analysis of covariance (ANCOVA) model was used to estimate the mean difference in the timeadjusted Area Under Curve (AUC) between the two treatment groups, with covariates for baseline scores and stratification factors. To test the treatment effect, a mixed linear model (random coefficient model) was used for the EQ-5D VAS score. Statistical tests were performed with a 2 sided type I error of 5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.978, 95% CI 2-sided [1.797 to 4.159]

6. Other Pre Specified Outcome: Patient Reported Outcomes: Functional Assessment of Cancer Therapy (FACT)- Hepatobiliary Subscale (HEP) Score
Description: The FACT-HEP is a 45 item, self-administered, multi-dimensional, psychometrically sound questionnaire used extensively in oncology clinical trials. FACT-HEP consisted of five subscales: Physical Well-Being (PWB), Social Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB), and Hepatobiliary Cancer Subscale (HCS). The PWB, FWB, SWB and EWB were summed to form the FACTGeneral (FACT-G) total score. The FACT-G and HCS scores were summed to form the FACT-HEP total score. FACT-HEP scores ranged from 0 to 180 and the higher scores represented a better quality of life. Subjects responded to each item on a 5-point Likert-type scale ranging from 0 (not at all) to 4 (very much). The minimally important difference (MID) for the FACT-Hep total score was in the range of 8 to 9. The results on the ANCOVA analysis of time-adjusted AUC for the FACT-HEP score were reported.
Time Frame: Cycle (C) Day (D)1, C2D1, C3D1 and subsequent cycles up to C18, end of intervention visit
Population: FAS included participants who were randomized to study treatments.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Unit on a scale | 138.7 [135.9 to 141.5] | 143.79 [141.1 to 146.5]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; An ANCOVA model was used to estimate the mean difference in the timeadjusted AUC between the two treatment groups, with covariates for baseline scores and stratification factors. To test the treatment effect, a mixed linear model (random coefficient model) was used for the FACT-HEP score. Statistical tests were performed with a 2 sided type I error of 5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [3.5 to 6.7]

7. Other Pre Specified Outcome: Patient Reported Outcomes: Functional Assessment of Cancer Therapy (FACT)- General (G) Total Score
Description: The PWB, FWB, SWB and EWB were summed to form the FACT-G total score. Subjects responded to each item on a 5-point Likert-type scale ranging from 0 (not at all) to 4 (very much). FACT-G scores ranged from 0 to 108 and the higher scores represented a better quality of life. The MID for the FACT-G total score was in the range of 6 to 7. The results on the ANCOVA analysis of time-adjusted AUC for the FACT-G score were reported.
Time Frame: Cycle (C) Day (D)1, C2D1, C3D1 and subsequent cycles up to C18, end of intervention visit
Population: FAS included participants who were randomized to study treatments.
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 556 | 558
Unit on a scale | 80.46 [78.6 to 82.3] | 82.95 [81.1 to 84.8]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; An ANCOVA model was used to estimate the mean difference in the timeadjusted AUC between the two treatment groups, with covariates for baseline scores and stratification factors. To test the treatment effect, a mixed linear model (random coefficient model) was used for the FACT-G score. Statistical tests were performed with a 2 sided type I error of 5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [1.4 to 3.6]

8. Other Pre Specified Outcome: The Correlation Between Plasma Biomarker Levels at Baseline With RFS to Determine Prognostic Value of Biomarkers - ANG-2
Description: Biomarker was analyzed at baseline [i.e., before treatment] as a dichotomized variable based on median biomarker levels, and dichotomized into "high" and "low" groups using an optimal max chi cut-off approach - not per intervention. As such, results were analyzed according to this stratification. Max-chi square methodology was used to search for the optimal cut point for dichotomization of each plasma biomarker and Kaplan-Meier curves were generated using the optimal cut point for each possible association examined. These biomarker analyses were retrospective and exploratory and of signal generating nature only.
Time Frame: At Baseline
Population: Plasma biomarker analysis was done in 858 (77%) of the all enrolled subjects.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- ANG-2 High Expression Group: ANG-2 high expression group included participants with the ANG-2 expression higher than 4009.765 pg/mL.
- ANG-2 Low Expression Group: ANG-2 low expression group included participants with the ANG-2 expression lower than 4009.765 pg/mL.
Arm/Group | ANG-2 High Expression Group | ANG-2 Low Expression Group
Number analyzed (Participants) | 258 | 600
Days | 588 [344 to 839] | 1260 [1026 to NA] — Value cannot be estimated due to censored data.
Statistical Analysis 1: Comparison: ANG-2 High Expression Group vs ANG-2 Low Expression Group; Test type: Superiority or Other; Hazard Ratio (HR) = 1.562, 95% CI 2-sided [1.241 to 1.965] — Significance of the biomarker main effect (RFS) and its corresponding hazard ratio estimate (HR) with 95% CI were reported. HR was expressed as high/low biomarker levels

9. Other Pre Specified Outcome: The Correlation Between Plasma Biomarker Levels at Baseline With RFS to Determine Prognostic Value of Biomarkers - AFP
Description: as for outcome 8
Time Frame: At Baseline
Population: Plasma biomarker analysis was done in 858 (77%) of the all enrolled subjects.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- AFP High Expression Group: AFP high expression group included participants with the AFP expression higher than 3.899 ng/mL.
- AFP Low Expression Group: AFP low expression group included participants with the AFP expression lower than 3.899 ng/mL.
Arm/Group | AFP High Expression Group | AFP Low Expression Group
Number analyzed (Participants) | 333 | 525
Days | 668 [420 to 924] | 1267 [1094 to NA] — Value cannot be estimated due to censored data.
Statistical Analysis 1: Comparison: AFP High Expression Group vs AFP Low Expression Group; Test type: Superiority or Other; Hazard Ratio (HR) = 1.747, 95% CI 2-sided [1.407 to 2.170] — [estimate comment as in outcome 8, analysis 1]

10. Other Pre Specified Outcome: The Correlation Between Plasma Biomarker Levels at Baseline With RFS to Determine Prognostic Value of Biomarkers - MET
Description: as for outcome 8
Time Frame: At Baseline
Population: Plasma biomarker analysis was done in 858 (77%) of the all enrolled subjects.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- MET High Expression Group: MET high expression group included participants with the MET expression higher than 182.444 ng/mL.
- MET Low Expression Group: MET low expression group included participants with the MET expression lower than 182.444 ng/mL.
Arm/Group | MET High Expression Group | MET Low Expression Group
Number analyzed (Participants) | 632 | 226
Days | 841 [675 to 1008] | NA [1262 to NA] — Value cannot be estimated due to censored data.
Statistical Analysis 1: Comparison: MET High Expression Group vs MET Low Expression Group; Test type: Superiority or Other; Hazard Ratio (HR) = 1.560, 95% CI 2-sided [1.206 to 2.018] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: From the date of signing informed consent up to 30 days post-treatment discontinuation
Description: In the safety analysis set (SAF), subjects were analyzed as treated but not randomized, therefore, few subjects in the placebo group of the full analysis set were switched to the sorafenib group of the SAF. Hence, SAF for safety analyses comprised of 548 subjects in the placebo group and 559 subjects in the sorafenib group.
Groups:
- Placebo: Subjects received 2 tablets of placebo orally twice daily.
- Sorafenib (Nexavar, BAY43-9006): Subjects received 2 tablets of Sorafenib [2*200 milligram (mg)] orally twice daily.
Arm/Group | Placebo | Sorafenib (Nexavar, BAY43-9006)
Serious Adverse Events (participants affected / at risk) | 230/548 | 228/559
Other Adverse Events (participants affected / at risk) | 360 | 522
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=548) | Sorafenib (Nexavar, BAY43-9006) (N=559)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (3)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (2) | 1 (2)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (5)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (5)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 4 (6)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (4)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 2 (5)
Large intestine perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (6)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 2 (3) | 2 (2)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 (5) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (4)
Multi-organ failure (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Coronary artery restenosis (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary fistula (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 4 (9)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (5)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (3)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 3 (4)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (2) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (2)
Peritonitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Superinfection (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 3 (4) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Bone formation increased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (16) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 4 (8)
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 130 (154) | 82 (98)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (4)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 3 (7)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (2)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 1 (2)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (4) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinusitis noninfective (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Incisional hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Neoplasm prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Removal of foreign body from gastrointestinal tract (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Inferior vena caval occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 1 (1)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Sorafenib (Nexavar, BAY43-9006)
Thrombocytopenia (Blood and lymphatic system disorders) | 14/548 (97) | 29/559 (217)
Abdominal pain (Gastrointestinal disorders) | 46/548 (115) | 55/559 (156)
Abdominal pain upper (Gastrointestinal disorders) | 14/548 (36) | 28/559 (75)
Ascites (Gastrointestinal disorders) | 19/548 (67) | 39/559 (145)
Constipation (Gastrointestinal disorders) | 36/548 (122) | 41/559 (105)
Diarrhoea (Gastrointestinal disorders) | 64/548 (186) | 242/559 (1201)
Dyspepsia (Gastrointestinal disorders) | 30/548 (125) | 20/559 (112)
Nausea (Gastrointestinal disorders) | 24/548 (45) | 50/559 (119)
Fatigue (General disorders) | 66/548 (300) | 83/559 (315)
Pyrexia (General disorders) | 24/548 (32) | 33/559 (39)
Nasopharyngitis (Infections and infestations) | 38/548 (69) | 30/559 (66)
Alanine aminotransferase increased (Investigations) | 38/548 (177) | 54/559 (251)
Aspartate aminotransferase increased (Investigations) | 35/548 (188) | 51/559 (226)
Platelet count decreased (Investigations) | 26/548 (202) | 48/559 (300)
Weight decreased (Investigations) | 13/548 (41) | 60/559 (254)
Weight increased (Investigations) | 42/548 (310) | 14/559 (68)
Decreased appetite (Metabolism and nutrition disorders) | 18/548 (52) | 40/559 (104)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30/548 (139) | 34/559 (162)
Back pain (Musculoskeletal and connective tissue disorders) | 37/548 (192) | 43/559 (152)
Headache (Nervous system disorders) | 33/548 (108) | 40/559 (111)
Insomnia (Psychiatric disorders) | 31/548 (178) | 24/559 (111)
Cough (Respiratory, thoracic and mediastinal disorders) | 44/548 (116) | 30/559 (76)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3/548 (7) | 41/559 (133)
Alopecia (Skin and subcutaneous tissue disorders) | 18/548 (65) | 187/559 (750)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 27/548 (139) | 390/559 (2196)
Pruritus (Skin and subcutaneous tissue disorders) | 58/548 (263) | 47/559 (133)
Rash (Skin and subcutaneous tissue disorders) | 45/548 (126) | 95/559 (296)
Hypertension (Vascular disorders) | 65/548 (331) | 142/559 (869)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days